CLINICAL TRIAL: NCT03099590
Title: Alkontrol-herbal (Isoflavone) Effects on Alcohol Drinking in an Outpatient Setting
Brief Title: Alkontrol-herbal Effects on Alcohol Drinking
Acronym: Alkontrol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Scott Lukas, Director - McLean Imaging Center, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017P000109
Record Dates: First submitted 2017-03-11; First posted 2017-04-04 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Alcohol Drinking; Alcohol Use Disorder; Alcohol Abstinence
MeSH Terms: conditions — Alcohol Drinking; Alcoholism; Alcohol Abstinence | interventions — puerarin

STUDY DESIGN:
Intervention Model Description: Half of the enrolled subjects will receive treatment with Alkontrol-herbal, kudzu extract, and half will receive a placebo control.
Who Masked: Participant, Care Provider
Masking Description: Neither the participants nor the study personnel providing the care/assessments will know whether the treatment received is active or placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment, Alkontrol-herbal (Experimental): Alkontrol-herbal, a kudzu extract which contains 19% puerarin, 4% daidzin and 2% daidzein, so each capsule contains a total of 25% active isoflavones or 125 mg.
  Interventions: Dietary Supplement: kudzu extract, puerarin
- Placebo Control (Placebo Comparator): Matched dextran containing capsules will serve as placebo.
  Interventions: Dietary Supplement: Placebo control

INTERVENTIONS:
Dietary Supplement: kudzu extract, puerarin — Capsules containing 500 mg of a crude kudzu extract (NPI-031, Alkontrol-herbal; Natural Pharmacia International, Burlington, MA) will be used, containing 19% puerarin, 4% daidzin and 2% daidzein, so each capsule contains a total of 25% active isoflavones or 125 mg.
  Other Names: Alkontrol-herbal
  Arms: Active Treatment, Alkontrol-herbal
Dietary Supplement: Placebo control — Matched sugar beet placebo capsules will serve as placebo.
  Arms: Placebo Control

SUMMARY:
Participants will enroll in a 14-week study (2 weeks of baseline, 8 weeks of treatment, and 4 weeks of follow-up) investigating the impact that Alkontrol-herbal (Isoflavone; Kudzu) has on alcohol intake in a population seeking treatment for an alcohol use disorder.

DETAILED DESCRIPTION:
Over the past 15 years, the Behavioral Psychopharmacology Research Lab at McLean Hospital has extensively studied kudzu extract and demonstrated its safety and efficacy in healthy control subjects as well as in heavy binge drinkers. The relative success of our recent outpatient trial of kudzu extract demonstrated a modest decrease in drinking, reduction in the number of heavy drinking days, and significant increase in the number of days abstinent. This suggests that Alkontrol-herbal, kudzu extract, may be a useful adjunct in treating alcohol use disorders.

Participants will enroll in a 14-week study (2 weeks of baseline, 8 weeks of treatment, and 4 weeks of follow-up) investigating the impact that Alkontrol-herbal has on alcohol intake in a population (age 21-60 years) seeking treatment for an alcohol use disorder. Participants will take 500 mg of a crude kudzu extract (NPI-031, Alkontrol-herbal; Natural Pharmacia International, Burlington, MA) t.i.d.; matched sugar beet placebo capsules will serve as placebo. Subjects will come to the lab three times a week to provide urine samples that can be tested for medication compliance through a biochemical marker, acetazolamide, included in the medication capsules. Participants will record their alcohol intake through daily diaries and a wrist actigraphy device, which will also monitor their sleep/wake activity.

ELIGIBILITY:
Inclusion Criteria:

* Subject can understand and comply with the protocol
* Good physical and mental health (normal physical exam, ECG, blood and urine chemistries, including absence of history or laboratory evidence of diabetes)
* Body Mass Index between 18-30, inclusive
* Age 21-60 years (age will be verified by driver's license or other valid form of identification)
* Meet criteria for current Moderate or Severe (4+ symptoms) Alcohol Use Disorder per the DSM-5; If attending a self-help treatment group (e.g., AA) at time of the screening visit, subject must agree to continue attending these groups for the duration of the study
* Seeking treatment for an Alcohol Use Disorder
* Drink 20-35 (or more) drink per week
* Report drinking on 80% of days in the past 90 days
* Have a stable living situation with current postal address

Exclusion Criteria:

* Subject meets DSM-5 criteria for major depression and/or bipolar disorder, and is not medically, pharmacologically, or clinically stable. Subjects who currently meet criteria for minor depression or bipolar disorder and have been clinically stable (including medications) for the past 2 months may participate in the study, at the investigator's discretion
* Concurrent diagnosis of any other Axis I disorder, including any substance use disorder besides alcohol use disorder Maintained on an antipsychotic or anti-seizure medication; Current prescription for benzodiazepines
* Presence of neurological, infectious, or neoplastic disease or a chronic medical disorder
* Tobacco use greater than 10 cigarettes per day
* Currently abstaining from consuming alcoholic beverages longer than 10 days
* History of major head trauma resulting in cognitive impairment or history of seizure disorder
* Heavy caffeine use (greater than 500 mg on a regular, daily basis)
* Subject has active hepatitis and/or aspartate aminotransferase (AST), alanine aminotransferase (ALT) > 3x the upper limit of normal
* For female volunteers, a positive pregnancy test (female subjects must agree to an approved method of contraception for the duration of the study)

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
percent days abstinent | change from baseline to post 8 weeks of treatment
  percent days abstinent from alcohol
drinks/day | change from baseline to post 8 weeks of treatment
  number of alcoholic drinks/day reported
number (or percent) of heavy drinking days | change from baseline to post 8 weeks of treatment
  number (or percent) of heavy drinking days
percent days abstinent | change from baseline to 4 weeks follow-up post-treatment
  percent days abstinent from alcohol
drinks/day | change from baseline to 4 weeks follow-up post-treatment
  number of alcoholic drinks/day reported
number (or percent) of heavy drinking days | change from baseline to 4 weeks follow-up post-treatment
  number (or percent) of heavy drinking days

CONTACTS AND LOCATIONS:
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No